CLINICAL TRIAL: NCT05936268
Title: A Randomized, Open Lable, Multi-center, Active Competitor Phase 2 Study for Evaluating Efficacy and Safety of Genakumab for Injection as First Line Therapy in Patients With Gout Flare
Brief Title: Safety and Efficacy of Genakumab for Injection in Patients With Gout Flare
Acronym: Gensci 048-203
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Collaborators: Huashan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GenSci048-203
Record Dates: First submitted 2023-06-30; First posted 2023-07-07 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Acute Gout; Gout Flare
Keywords: Acute gout; Gout flare
MeSH Terms: interventions — Injections; Colchicine

STUDY DESIGN:
Intervention Model Description: Acute gout patients with gout flare Group A: Genakumab 200mg single injection;Group B: Etoricorxib 120mg qd po.(until remission or intorlerance, no longer than 8 days)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Genacumab group (Experimental): Genakumab 200mg single injection
  Interventions: Drug: Genakumab for injection
- cholchicine group (Active Comparator): Colchicine 0.5mg qd po.for 12 weeks
  Interventions: Drug: Colchicine

INTERVENTIONS:
Drug: Genakumab for injection — 150 mg/1ml/bottle
  Arms: Genacumab group
Drug: Colchicine — 0.5mg/table
  Arms: cholchicine group

SUMMARY:
To evaluate the safety and efficacy of Genakumab for Injection in patients with gout flare as a first line therapy

DETAILED DESCRIPTION:
Phase 2， randomized, open lable, multi-center, active controlled study. Patients are randomized to Genakumab 200mg single injection group or Etoricorxib 120mg qd po.(until remission or intorlerance, no longer than 8 days) group.

ELIGIBILITY:
1. Male or female, 18 years ≤ age ≤ 75 years;
2. BMI ≤ 40kg/m2
3. Meeting ACR 2015 preliminary criteria for the classification of acute arthritis of primary gout;
4. Start of acute gout flare within 3 days prior to enrolled;
5. History of ≥2 gout flare within 12 months prior to study start;
6. Baseline pain intensity ≥ 50mm on the 0-100mm visual analog scale(VAS)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2023-07-21 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
72hours target joint VAS change from baseline | 72h±2h
  72hours target joint VAS change from baseline

SECONDARY OUTCOMES:
Pain intensity | 6hours, 24hours, 48hours, 72hours, Day 8,
  target joint VAS Target joint VAS change from baseline Time to first VAS<=50% baseline VAS Time to first VAS<=30mm Time to first VAS<=10mm
Recurrence of flare | 12 weeks after the last dose
  Proportion of patients who have at least 1 flare Time to first flare
Safety outcome | 12weeks
  AE, laboratory examination, ECG, vital signs and physical examination
immunogenic outcome | 12 weeks after the last dose
  The incidence of anti-drug antibodies (ADA) and the incidence of neutralizing antibody

CONTACTS AND LOCATIONS:
Overall Officials: Hejian Zou, Principal Investigator — Fudan University Affiliated Huashan Hospital
Locations (1):
- Fudan University Affiliated Huashan Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Kong N, Xue Y, Mao L, Qian L, Guo H, Hu J, Yuan F, Li R, Duan X, Yu J, Gou W, Yang L, Wei H, Li R, Xu Q, Luo T, Zhang X, Zou H. Efficacy and Safety of Firsekibart Compared to Etoricoxib for Gout Flares: A Phase 2, Multicenter, Open-label, Active-controlled, Randomized Non-inferiority Trial. Rheumatol Ther. 2025 Oct;12(5):975-990. doi: 10.1007/s40744-025-00790-6. Epub 2025 Aug 20. PMID 40833487